CLINICAL TRIAL: NCT04772131
Title: Prospective, Post-market Study of the Desara® One Single Incision Sling vs. Desara® Blue Sling Implanted Via the Transobturator Route for the Treatment of Women With Stress Urinary Incontinence
Brief Title: Desara ® One Single Incision Sling 522 Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Caldera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PS200005
Record Dates: First submitted 2021-02-05; First posted 2021-02-26 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Stress Urinary Incontinence
Keywords: stress urinary incontinence; female stress urinary incontinence; single incision sling; transobturator sling; Desara® One; Desara® Blue
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Adult female subjects, who in the opinion of their physician require surgical treatment or who have already been diagnosed with stress urinary incontinence, will be eligible for study participation. Subjects who provide informed consent will undergo screening and baseline assessments. Subjects who successfully meet the study's inclusion and exclusion criteria will be eligible to undergo a Desara SIS or Desara Blue implant procedure, with subsequent follow-up assessments. The choice of implant, Desara One or Desara Blue, will be determined by the investigator based upon patient pathology and surgical preference.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Desara® One (Experimental): Single Incision Sling
  Interventions: Device: Desara® One Single Incision Sling
- Desara® Blue (Active Comparator): Transobturator Sling
  Interventions: Device: Desara® Blue Transobturator Sling

INTERVENTIONS:
Device: Desara® One Single Incision Sling — Single incision sling
  Arms: Desara® One
Device: Desara® Blue Transobturator Sling — Standard mid-urethral sling
  Arms: Desara® Blue

SUMMARY:
A post-market study to compare the safety and effectiveness of the Desara® One Single Incision Sling (SIS), when compared to that of an FDA cleared transobturator sling over a period of 36 months.

DETAILED DESCRIPTION:
This study is a prospective, non-randomized, parallel cohort, multi-center study of Desara® One single incision sling (SIS) compared to Desara® Blue sling systems implanted via the transobturator-route (TOR) for the treatment of women with stress urinary incontinence (SUI). The study will compare results from SIS patients (N=150) and TOR patients (N=150) at up to 40 sites for a total period of 36 months, with follow-up visits at 2 and 6 weeks, 6, 12, 18, 24 and 36 months. This study will enroll adult females who are clinically indicated for a mid-urethral implant for the treatment of female stress urinary incontinence (SUI) resulting from urethral hypermobility and/or intrinsic sphincter deficiency (ISD).

ELIGIBILITY:
Inclusion Criteria:

1. Female ≥ 18 of age.
2. Subject agrees that she is willing and able to return for all study related procedures and evaluations.
3. Subject has provided signed informed consent.
4. Subject has stress urinary incontinence (SUI) confirmed by either supine or standing cough stress test (CST) with bladder pre-fill to subjective fullness with 200-300 mL, or with bladder fullness confirmed via ultrasound.
5. Subject has confirmed stress incontinence greater than urge incontinence per MESA questionnaire.
6. Subject no longer has childbearing capacity or has a negative pregnancy test and has decided to cease childbearing. Childbearing capacity to be confirmed by documented history of:

   1. A hysterectomy or
   2. Tubal ligation or
   3. Is otherwise incapable of pregnancy or has
   4. Negative pregnancy test prior to study entry and has decided to cease childbearing
7. Subject has been offered and either failed or refused alternative non-invasive SUI treatment options and has elected to proceed with a surgical intervention.
8. Subject is eligible to undergo laparoscopic/robotic (with or without mesh) or vaginal (with or without mesh) apical, anterior or posterior prolapse concomitant surgical repair procedures (non-mesh).

Exclusion criteria:

1. Subject reports baseline pelvic pain ≥ 2 on 10 point Numeric Rating Scale (NRS).
2. Subject has a known neurological disease (with or without signs/symptoms of neurogenic bladder).
3. Subject has known pre-existing pain syndrome and/or has been evaluated by an interventional pain management physician.
4. Subject has a history of chronic opioid, or narcotic use for:

   1. pain or
   2. any other specified reason
5. Subject is on anti-coagulation therapy that cannot be suspended or adjusted for a minimum of 24-48 hours prior to planned sling implantation surgery.
6. Subject is on chronic (> 3 months) systemic steroid treatment (except for inhalational use as indicated for pulmonary conditions).
7. Subject has uncontrolled diabetes defined as A1c ≥ 7% or fasting serum glucose > 130mg/dl at screening/baseline.
8. Subject has an active lesion or skin infection of the perineum, urethra, or vagina as noted per visual pelvic exam.
9. Subject has active UTI which requires treatment, as determined by the Investigator.
10. Subject has pattern of recurrent UTIs, defined as ≥ 3 culture-proven UTIs during the 6-month period prior to surgery.
11. Subject has a urethral obstruction or other anatomic defects of the urethra (inclusive of urethral diverticulum or stricture or bladder neck contracture).
12. The subject has had:

    1. any prior surgical stress urinary incontinence treatment or
    2. any prior surgery on their urethra or
    3. any prior surgery to distal anterior vaginal wall, including fistula repair or prior cystocele repair
    4. any previous pelvic floor mesh use or complication
13. Subject has any of the following confounding conditions:

    1. bladder stones or tumors
    2. pathology that in the opinion of the Investigator would compromise implant placement
    3. pathology that would limit pelvic blood supply
    4. pathology that would require chemotherapy and systemic use of immunosuppressants
14. Subject has abnormal bladder capacity <300 mL.
15. Subject has a post void residual volume ≥ 150 mL on two different measurements. (Prolapse reduction during PVR measurement is only allowed if a prolapse repair will be performed concomitantly with the sling implantation)
16. Subject has had previous radiation therapy or brachytherapy to the pelvis.
17. Subject is enrolled in a concurrent clinical trial of any treatment (drug or device) that could affect continence function, interfere with clinical outcomes, or impact analysis of this device.
18. Subject has known reaction, sensitivity or allergy to polypropylene.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Success rate of negative standing cough stress test (CST) | 36 months
  Negative standing cough stress test (CST) with bladder pre-fill to subjective fullness with 200-300 mL, or with bladder fullness confirmed via ultrasound, evaluated at the 36-month post-implant follow-up visit. The success rate is defined as the proportion of subjects with a negative CST at the 36-month post-implant follow-up
Device and Procedure-related serious adverse events | 36 months
  * Device- and/or procedure-related adverse event rates at the post-implant follow-up visits
  * Revision/re-surgery rates at post-implant follow-up visits
  * Device and/or procedure-related serious adverse events

SECONDARY OUTCOMES:
Composite outcome success rates | 6 weeks, 6, 12, 18, 24, 36 months
  Defined by the primary effectiveness endpoint and subjective measure of Improvement in the Patient Global Impression of Improvement (PGI-I) index for incontinence post-implant
Sexual Function Assessment | 6 weeks, 6, 12, 18, 24, 36 months
  Use of PISQ-12: Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire to assess subject changes in sexual function
Improvement in Incontinence | 6 weeks, 6, 12, 18, 24, 36 months
  Use of PGI-I: Patients Global Impression of Improvement index for incontinence to assess subject improvement post-implant
Improvement in Urinary Symptoms | 6 weeks, 6, 12, 18, 24, 36 months
  Use of IIQ-7: Incontinence Impact Questionnaire, Short Form and ICIQ-UI: International Consultation on Incontinence Questionnaire-Urinary Incontinence to assess improvement in urinary symptoms post-implant
Improvement in Urge and Stress Incontinence | 6 weeks, 6, 12, 18, 24, 36 months
  Use of UDI-6 SF: Urinary Distress Inventory, Short Form to assess subject improvement in urge and stress incontinence post-implant
Subject pain assessment | 6 weeks, 6, 12, 18, 24, 36 months
  Use of Numeric Rating 10-point scale (NRS) to assess post-operative pain. Pain scale is 0= no pain to 10 = worst pain
Time to void post-implant | 6 weeks, 6, 12, 18, 24, 36 months
  Perform a standard post void residual test to confirm that the subject's residual urine volume is ≥150 mL

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Valley Urogynecology Associates, Inc., Phoenix, Arizona
  - University of Arizona College of Medicine, Tucson, Arizona
  - Urological Research Center Corp, Hialeah, Florida
  - Women's Health Care Associates P.A. dba Rosemark Women Care Specialists, Idaho Falls, Idaho
  - CMB Research, LLC, Newburgh, Indiana
  - University of Louisville, Louisville, Kentucky
  - Mt. Auburn Hospital Division of Urogynecology, Cambridge, Massachusetts
  - Specialty Clinical Research of St. Louis, LLC, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - University of New Mexico, Albuquerque, New Mexico
  - Novant Health Urogynecology, Charlotte, North Carolina
  - The Lindner Research Center at The Christ Hospital, Cincinnati, Ohio
  - Center for Total Women's Health, Lansdale, Pennsylvania
  - Center for Pelvic Health, Franklin, Tennessee
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No